CLINICAL TRIAL: NCT05883995
Title: Avis-PHAGEinLYON Clinic
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 23-5092
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Bone Infection
Keywords: bacteriophage; medical advice

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Phage therapy requests — Quantification of phage therapy requests received at the Hospices Civils de Lyon from 2015 to 2028

SUMMARY:
Avis-PHAGEinLYON Clinic study is a single site non-interventional retrospective and prospective study, initiated by the Hospices Civils de Lyon. Population targeted are patients referred to the Hospices Civils de Lyon for a medical advice for a phage therapy from 2015 to 2028. The primary objective is to quantify the phage therapy requests received at the Hospices Civils de Lyon. 1500 patients will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* - Patient referred to the Hospices Civils de Lyon for a phage therapy request from 01/01/2015 to 01/01/2028.
* Avis-PHAGEinLYON clinic study information notice provided to the patient

Exclusion Criteria:

* - Opposition of trial participant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1500 patients with severe infection treated with phagotherapy will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of phage therapy requests | at inclusion
  Number of phage therapy requests received at the Hospices Civils de Lyon from 2015 to 2028 per year and per month.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Référence des Infections Ostéo-Articulaires complexes (CRIOAc) - Hôpital de la Croix-Rousse, Lyon, France

REFERENCES:
- [Derived] Ferry T, Bouar ML, Briot T, Roussel-Gaillard T, Perpoint T, Roux S, Ader F, Valour F, Kassai B, Boussaha I, Ndiaye M, Craighero F, Javaux C, Lustig S, Batailler C; PHAGEinLYON Clinic Study Group. Access to phage therapy at Hospices Civils de Lyon in 2022: Implementation of the PHAGEinLYON Clinic programme. Int J Antimicrob Agents. 2024 Dec;64(6):107372. doi: 10.1016/j.ijantimicag.2024.107372. Epub 2024 Nov 2. PMID 39491599